CLINICAL TRIAL: NCT02702011
Title: A Phase II, Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Once Daily, Oral Doses of Empagliflozin as Adjunctive to Insulin Therapy for 28 Days in Japanese Patients With Type 1 Diabetes Mellitus
Brief Title: Empa Add on to Insulin in Japanese Patient With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.113
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Results first posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — empagliflozin

ARMS (4):
- empagliflozin low dose (Experimental)
  Interventions: Drug: empagliflozin low dose
- empagliflozin medium dose (Experimental)
  Interventions: Drug: empagliflozin medium dose
- empagliflozin high dose (Experimental)
  Interventions: Drug: empagliflozin high dose
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: empagliflozin medium dose
  Arms: empagliflozin medium dose
Drug: empagliflozin low dose
  Arms: empagliflozin low dose
Drug: empagliflozin high dose
  Arms: empagliflozin high dose
Drug: placebo
  Arms: placebo

SUMMARY:
To assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of once daily oral doses of empagliflozin in Japanese patients with type 1 diabetes mellitus as adjunctive therapy to insulin.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent by the date of Visit 1 (screening) in accordance with Good Clinical Practice (GCP) and local legislation
* Japanese male or female patient receiving insulin for treatment of documented diagnosis of type 1 diabetes mellitus (T1DM) for at least 1 year at the time of Visit 1 (screening).
* Fasting C-peptide value of < 0.6 ng/mL at Visit 2 (placebo run-in) measured by the central laboratory
* Use of, and be willing, based on the investigator's judgment, to continue throughout the duration of the trial Multiple daily injection(MDI) of insulin consisting of at least 1 basal insulin injection and at least 3 daily bolus injections The total daily insulin dose must be>=0.3 U/kg and <=1.5 U/kg at Visit 1 (screening)
* HbA1c of 7.5% to 10.0% at Visit 1 (screening) measured by the central laboratory and provided that the patients HbA1c does not increase by > 0.5% within 3 months before Visit 1 (screening)
* Based on the investigator's judgment, patient must have a good understanding of his/her disease and how to manage it, and be willing and capable of performing the following study assessments (assessed at Visits 1 to 3 and just before randomization)
* patient-led management and adjustment of insulin therapy
* reliable approach to insulin dose adjustment for meals, such as carbohydrate counting
* reliable and regular home-based blood glucose monitoring
* recognize the symptoms of DKA (Diabetic Ketoacidosis), and reliably monitor for ketones
* implementation of an established "sick day" management regimen
* Age >=20 years and <=65 years at Visit 1 (screening)
* Body mass index (BMI) >=18.5 kg/m2 and<=35.0 kg/m2 at Visit 1 (screening)
* Estimated glomerular filtration rate (eGFR) >=60 mL/min/1.73m² and <=150 mL/min/1.73m² as calculated by Japanese equation based on creatinine measured by the central laboratory at Visit 1 (screening)
* Compliance with trial drug administration must be between 80% and 120% during the placebo run-in period, to be judged at Visit 4 and before randomization

Exclusion criteria:

* History of T2DM (Type 2 Diabetes Mellitus), maturity onset diabetes of the young (MODY), pancreatic surgery or chronic pancreatitis
* Pancreas, pancreatic islet cells or renal transplant recipient
* T1DM treatment with any other anti-hyperglycaemic drug (e.g., metformin, alpha-glycosidase inhibitors, glucagon-like-peptide 1 (GLP-1) receptor agonists, SGLT-2 (Sodium-Glucose co-transporter-2) inhibitors, pramlintide, inhaled insulin, pre-mixed insulins, etc.) within 3 months except subcutaneous basal and bolus insulin before Visit 1 (screening) or any history of clinically relevant hypersensitivity according to the investigator's judgment
* Occurrence of severe hypoglycemia involving coma and/or seizure that required hospitalization or hypoglycemia-related treatment by an emergency physician or paramedic within 3 months before Visit 1 (screening)
* Occurrence of DKA within 3 months before Visit 1 (screening) and until randomization at Visit 4 (Day 1)
* Irregular sleep/wake cycle (e.g., patients who habitually sleep during the day and work during the night) based on the investigator's judgment
* Acute coronary syndrome (non-STEMI, STEMI, and unstable angina pectoris), stroke or transient ischemic attack within 3 months before Visit 1 (screening)
* Diagnosis of severe gastro paresis based on investigator's judgment
* Diagnosis of brittle diabetes based on the investigator's judgment
* Indication of liver impairment, defined by serum levels of either alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase above 3 x upper limit of normal (ULN) at Visit 1 (screening) as measured by the central laboratory
* Eating disorders such as bulimia or anorexia nervosa
* Treatment with anti-obesity drugs (e.g., Mazindol), surgery or aggressive diet regimen leading to unstable body weight (based on the investigator's judgment) 3 months before Visit 1 (screening) and until randomization
* Treatment with systemic corticosteroids or planned initiation of such therapy at Visit 1 (screening). Inhaled use of corticosteroids (e.g., for asthma/chronic obstructive pulmonary disease) is acceptable
* Change in dose of thyroid hormones within 6 weeks before Visit 1 (screening) or planned change or initiation of such a therapy at Visit 1 (screening)
* Medical history of cancer or treatment for cancer in the last 5 years before Visit 1 (screening). Resected basal cell carcinoma considered cured is exempted
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells (e.g., malaria, babesiosis, hemolytic anemia) at Visit 1 (screening)
* Pre-menopausal women (last menstruation <=1 year before informed consent) who:
* are nursing or pregnant or
* are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, intra uterine devices/systems, oral contraceptives, complete sexual abstinence, double barrier method and vasectomized partner
* Alcohol or drug abuse within 3 months before Visit 1 (screening) that would interfere with trial participation based on the investigator's judgment
* Intake of an investigational drug in another trial within 30 days before Visit 1 (screening)
* Patient not able to understand and comply with study requirements based on the investigator's judgment
* Any other clinical condition that, based on investigator's judgment, would jeopardise patient safety or would affect the study outcome (e.g. immunocompromised patients who might be at higher risk of developing genital or mycotic infections, patients with chronic viral infections, etc.) during trial participation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-03-20 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2016-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Japan (4):
  - Souseikai Hakata Clinic, Fukuoka, Fukuoka
  - Nishikumamoto Hospital, Kumamoto, Kumamoto
  - Shinjuku Research Park Clinic, Tokyo, Shinjyuku-ku
  - SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku

REFERENCES:
- [Derived] Shimada A, Hanafusa T, Yasui A, Lee G, Taneda Y, Sarashina A, Shiki K, George J, Soleymanlou N, Marquard J. Empagliflozin as adjunct to insulin in Japanese participants with type 1 diabetes: Results of a 4-week, double-blind, randomized, placebo-controlled phase 2 trial. Diabetes Obes Metab. 2018 Sep;20(9):2190-2199. doi: 10.1111/dom.13351. Epub 2018 Jun 5. PMID 29766633

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral administration of matching placebo of 2.5 mg, 10 mg and 25 mg of empagliflozin film-coated tablets once daily during the 28 days randomized double-blinded treatment period.
- Empagliflozin 2.5 mg: Oral administration of 2.5 milligram (mg) of empagliflozin film-coated tablets once daily along with one matching placebo each of 10 mg and 25 mg of empagliflozin during the 28 days randomized double-blinded treatment period
- Empagliflozin 10 mg: Oral administration of 10 milligram (mg) of empagliflozin film-coated tablets once daily along with one matching placebo each of 2.5 mg and 25 mg of empagliflozin during the 28 days randomized double-blinded treatment period.
- Empagliflozin 25 mg: Oral administration of 25 milligram (mg) of empagliflozin film-coated tablets once daily along with one matching placebo each of 2.5 mg and 10 mg of empagliflozin during the 28 days randomized double-blinded treatment period.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Started | 11 (Started are the treated patients.) | 13 (Started are the treated patients.) | 12 (Started are the treated patients.) | 12 (Started are the treated patients.)
Completed | 11 | 12 | 12 | 12
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All patients randomised, treated with at least 1 dose of study drug, who had a baseline Urinary glucose excretion (UGE) (gram (g)/24 hour (h)) and a UGE (g/24 h) on Day 1 or Day 7.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg | Total
Number analyzed (Participants) | 11 | 13 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (11.7) | 44.2 (12.6) | 44.5 (11.8) | 46.6 (10.8) | 44.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 8 | 4 | 26
  Male | 5 | 5 | 4 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24 Hour UGE on Day 7
Description: Change from baseline in 24 hour urinary glucose excretion on Day 7 calculated as: UGE on Day 7 - UGE on baseline. Baseline is defined as the last observation prior to the first intake of any randomised trial medication.
Time Frame: Baseline and 7 days
Population: The primary analysis was performed on the FAS with last observation carried forward (LOCF) imputation.
Measure: Least Squares Mean (Standard Error); unit: gram per 24 hours (g/24 h)
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Number analyzed (Participants) | 11 | 13 | 12 | 12
gram per 24 hours (g/24 h) | -0.46 (7.96) | 64.63 (7.31) | 80.73 (7.68) | 97.64 (7.63)
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 2.5 mg; An analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline as a linear covariate was fitted to the change from baseline of 24 hour UGE (g/24h) on Day 7, where baseline refers to the last observation prior to the first intake of any randomised trial medication; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 65.10, 95% CI 2-sided [43.29 to 86.90], Standard Error of Mean 10.81 — Mean Difference was calculated as: (mean change from baseline in 24 hour UGE at Day 7 in Empagliflozin 2.5 mg group) - (mean change from baseline in 24 hour UGE at Day 7 in Placebo group)
Statistical Analysis 2: Comparison: Placebo vs Empagliflozin 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 81.19, 95% CI 2-sided [58.80 to 103.58], Standard Error of Mean 11.10 — Mean Difference was calculated as: (mean change from baseline in 24 hour UGE at Day 7 in Empagliflozin 10 mg group) - (mean change from baseline in 24 hour UGE at Day 7 in Placebo group)
Statistical Analysis 3: Comparison: Placebo vs Empagliflozin 25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 98.11, 95% CI 2-sided [75.91 to 120.31], Standard Error of Mean 11.01 — Mean Difference was calculated as: (mean change from baseline in 24 hour UGE at Day 7 in Empagliflozin 25 mg group) - (mean change from baseline in 24 hour UGE at Day 7 in Placebo group)

ADVERSE EVENTS:
Time Frame: From first drug administration till 7 days after last drug intake; up to 35 days
Description: Treated set (TS): This analysis set included all patients treated with at least one dose of randomised study drug.
Arm/Group | Placebo | Empagliflozin 2.5 mg | Empagliflozin 10 mg | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/11 | 12/13 | 12/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | Empagliflozin 2.5 mg (N=13) | Empagliflozin 10 mg (N=12) | Empagliflozin 25 mg (N=12)
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 12 | 12 | 12
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
A limitation of the current study is its short duration and small sample size. Another limitation of this study was that patients in the placebo group had to go through unnecessary dose adjustments of insulin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.